CLINICAL TRIAL: NCT03846765
Title: Influence of Continuous Administration of Phenylephrine Versus Dobutamine on Spinal Oxygen Saturation, Measured With Near-infrared Spectroscopy (NIRS).
Acronym: NIRS continu
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018/1510
Record Dates: First submitted 2019-02-15; First posted 2019-02-20 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Nfuence of Vasoactive Medication on Spinal Oxygenation
Keywords: spinal oxygenation; NIRS
MeSH Terms: interventions — Phenylephrine; Dobutamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phenylephrine continuous infusion (Experimental)
  Interventions: Drug: Phenylephrine
- Dobutamine continuous infusion (Experimental)
  Interventions: Drug: Dobutamine

INTERVENTIONS:
Drug: Phenylephrine — Phenylephrine will be administered continuously after intubation in order to maintain blood pressure in a range from MAPbaseline -20% to normal (preoperative) values (MAPbaseline). If MAP decreases to a value lower than MAPbaseline -20%, a higher dose of vasopressor will be administered. If MAP increases to a value above MAPbaseline, the dosing rate will be decreased.
  Phenylephrine will be started at 0,2 μg/kg/min and adjusted according to the patient's hemodynamic status. The dose will be adjusted to MAP during a 30-minute study period.
  Arms: Phenylephrine continuous infusion
Drug: Dobutamine — Dobutamine will be administered continuously after intubation in order to maintain blood pressure in a range from MAPbaseline -20% to normal (preoperative) values (MAPbaseline). If MAP decreases to a value lower than MAPbaseline -20%, a higher dose of vasopressor will be administered. If MAP increases to a value above MAPbaseline, the dosing rate will be decreased.
  Dobutamine will be started at 2 μg/kg/min; and adjusted according to the patient's hemodynamic status .The dose will be adjusted to MAP during a 30-minute study period.
  Arms: Dobutamine continuous infusion

SUMMARY:
To assess the effect of hemodynamic supportive medication on spinal vasculature, patients scheduled for arterial dilation of the lower limb were chosen as our study population. The spinal cord perfusion is not compromised in these patients, however, most patients suffer from hypotension during this kind of surgery, due to the non-invasive type of surgery and the vasodilating effects of the anesthetics. Therefore, continuous administration of vasoactive medication (phenylephrine or dobutamine) is often required in order to increase blood pressure.

The aim of our study is to evaluate the effect of a continuous administration of phenylephrine or dobutamine on the spinal oxygenation, assessed by NIRS.

DETAILED DESCRIPTION:
All patients receive standard anesthesia care during the surgical procedure. Before induction of anesthesia, baseline MAP will be defined and 6 additional sensors (stickers) will be applied to the back of the patient at three levels: 1 at the upper thoracic level(T3-T4), 2 at the lower thoracic level (T9-T10) and 2 at the lumbar region (L1-L2) and 1 on the deltoid muscle of the upper arm. Two sensors are routinely applied to the forehead to measure cerebral oxygenation and a BIS sensor is applied to measure depth of anesthesia. In all patients a non-invasive cardiac output monitor (Clearsight; EdwardsTM LifeScience, Irvine, CA, USA) is routinely used. This monitor provides a continuous arterial pressure waveform in a non-invasive way and facilitates continuous evaluation of blood pressure. Hereby, efficient adaptation of the administration of vasopressors is feasible. Through an intravenous line, anesthetics will be administered. Vasopressor agents will be administered through a dedicated second intravenous line. After induction of anesthesia, an endotracheal tube is placed.

A vasopressor agent will be administered continuously after intubation in order to maintain blood pressure in a range from MAPbaseline -20% to normal (preoperative) values (MAPbaseline). If MAP decreases to a value lower than MAPbaseline -20%, a higher dose of vasopressor will be administered. If MAP increases to a value above MAPbaseline, the dosing rate will be decreased. According to the group to which the patient has been randomized, phenylephrine or dobutamine will be administered and the dose will be adjusted to MAP during a 30-minute study period.

The total drug amount for phenylephrine and dobutamine will not exceed 5 mg, resp. 30 mg.

The study will be completed after 30 minutes of continuous medicamentous hemodynamic support administration (i.e. 30 minutes after intubation) or if administration of phenylephrine or dobutamine exceeds 1 µg/kg/min or 10 µg/kg/min, respectively.

If the administration of the study medication does not achieve the desired result, management of the hemodynamics will be left to the discretion of the attending anesthesiologist and the patient will be excluded from further data analysis.

The endovascular surgical procedure can start without delay and the duration of surgery will not be prolonged because of the measurements and blood pressure management

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18y
* Patient is scheduled for dilation of arterial blood vessels of the lower limb

Exclusion Criteria:

* Age < 18y
* BMI > 30
* severe valvular disease
* previous aortic surgery
* paraplegia/ paraparesis
* kidney replacement therapy
* pacemaker
* pregnancy
* lactating participants
* preoperative use of ACE inhibitors.
* No sinus rhythm on preoperative ECG or at induction of anesthesia (patients with a history of atrial fibrillation can be included if they have a sinus rhythm on their preoperative ECG)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2021-05-22 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Spinal oxygen saturation measured by NIRS | from intubation until 30 minutes after intubation
  Spinal oxygen saturation measured by NIRS

SECONDARY OUTCOMES:
Cerebral oxygen saturation | from intubation until 30 minutes after intubation
  Cerebral oxygen saturation measured by NIRS
Deltoid muscle oxygen saturation | from intubation until 30 minutes after intubation
  Deltoid muscle oxygen saturation measured by NIRS

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Vanpeteghem, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No